CLINICAL TRIAL: NCT00555516
Title: A Phase I/II Double-Blind, Randomized, Placebo-Control Pilot Study to Evaluate the Safety and Pharmacodynamic Activities of EW02 in Reducing Neutropenia Caused by Breast Cancer Chemotherapy
Brief Title: A Pilot Study to Evaluate the Safety and Activities of EW02 in Reducing Neutropenia Caused by Chemotherapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DOH96-TD-I-111-003
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2007-11-08 (Estimated); Status verified 2007-11

CONDITIONS: Breast Cancer; Chemotherapy; Neutropenia
Keywords: Breast Cancer、 Chemotherapy、 Neutropenia、WBC
MeSH Terms: conditions — Breast Neoplasms; Neutropenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 1. The chemotherapy regimen of group 1 is restricted to AC or CAF during the first cycle
  2. Group 1 will receive EW02 for 15 consecutive days during the second cycle
  3. will receive EW02 at 700mg tid/day for 15 consecutive days during the third cycle.
  Interventions: Other: EW02
- 2 (Placebo Comparator): 1. The chemotherapy regimen of group 2 is restricted to AC or CAF during the first cycle
  2. Group 2 will receive 15 consecutive days of Placebo
  3. Group 2 will receive EW02 at 700mg tid/day for 15 consecutive days during the third cycle
  Interventions: Other: EW02

INTERVENTIONS:
Other: EW02 — 1. Name: EW02
  2. Dosage form: capsule.
  3. Dose(s): 350mg per capsule, 2 capsule tid.
  4. Dosing schedule: 2 capsule tid; 15 days (D3 to D17) of EW02 or placebo in Cycles 2 and 3.

SUMMARY:
Study Hypothesis:

EW02 is a polysaccharide-enriched crude extract from black soybean (BS). BS has been used extensively by the Chinese as food or traditional Chinese medicine for hundreds of years. It has been used as monotherapy to treat Diabetes, menorrhagia and leukorrhea. In combination with others, BS has been used to treat chemotherapy-induced leukopenia on more than 300 pts. The daily doses were 15g bid to 50g tid for 21 days. Side effects were generally mild, including epigastric discomfort, numbness, insomnia, and dry mouth. Recently BS was found to promote myelopoiesis and inhibit tumor growth through immunomodulation. In vitro assays showed BS-PS can stimulate production of cytokines and increase blood progenitors. In vivo studies also demonstrated that BS-PS can reduce neutropenia in mice received 5-FU by stimulating myeloid colony formation. We hypothesize that EW02 can reduce neutropenia in cancer patients who receive chemotherapy without side effects.

DETAILED DESCRIPTION:
Study procedures:

This is a single-center, double-blind, placebo-controlled parallel, pilot study of oral EW02 in combination with chemotherapy, versus placebo in combination with chemotherapy in breast cancer patients as the primary phase (Cycle 1). The chemotherapy regimen is restricted to one of the following regimens: Doxorubicin + Cyclophosphamide (AC), or Doxorubicin+ Cyclophosphamide+5-FU (CAF) under standardized dosage. The WBC recovery time is similar between these two chemotherapy regimens due to the facts that doxorubicin and cyclophosphamide are overlapped and their dose in CAF is reduced. The principle investigator has clinical experiences that the neutropenia nadir and severity caused by these two regimens are almost the same. Nevertheless, pre-stratification by chemotherapy regimen (stratum AC versus stratum CAF) at randomization will be implemented so that equal sample size of two study products will be allocated under each stratum. It will involve 60 outpatients for breast cancer, who have previously demonstrated a fall unto 1,000 to 3,000/mm3 in WBC count, or unto 500 to 1,500/mm3 in ANC count, on Day 8 or Day 15, whilst on Cycle 1.

The second phase (Cycle 2): EW02 at 700mg tid daily versus placebo group are given at the beginning of Cycle 2 for 15 consecutive days. 60 subjects will be randomized 2:1 to two groups in pre-stratified permuted blocks of six with four subjects assigned to Group 1 (EW02) while two subjects assigned to Group 2 (Placebo). Group 1 will receive EW02 for 15 consecutive days during the second cycle and Group 2 will receive 15 consecutive days of Placebo.

The extension phase (Cycle 3): is designed to collect additional safety data and to ensure all the participants will have the opportunity to receive study drug. Thus, both groups will receive EW02 at 700mg tid/day for 15 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to inclusion in study
2. Pathologically confirmed breast cancer, whose CBC has shown ever dropped unto 1,000 to 3,000/mm3 in WBC count, or unto 500 to 1,500/mm3 in ANC count, on Day 8 or Day 15, whilst on Cycle 1 of current chemotherapy.
3. Age 20 - 70 years
4. Stage T 1-3, N 0-2, M0.
5. ECOG performance status of < 2
6. Chemotherapy regimen is restricted to one of the followings:

(1)Doxorubicin 60 mg/m2 + Cyclophosphamide 600 mg/m2(AC X 4cycles) or (2)Cyclophosphamide 500 mg/m2 + Doxorubicin 50 mg/m2 + 5-FU 500 mg/m2 (CAF X 6 cycles) 7.Laboratory test results within 30 days prior to study entry:

1. Hemoglobin 9.0 g/dL for men and 8.7 g/dL for women and platelet> 100,000/mm³ without the need for current, on-going use of erythropoietin or transfusion
2. Normal liver function (GOT < 1.5 x ULN)
3. Normal kidney function (Creatinine < 1.5 x ULN) and no dialysis. 8.Negative of mandatory pregnancy test for women subjects.

Exclusion Criteria:

1. Women under pregnancy or with positive result from mandatory pregnancy test or in lactating; women of child-bearing potential must use adequate contraception
2. Prior systemic therapy or radiotherapy for breast cancer
3. Known hypersensitivity to bean products
4. Serious medical or psychiatric illness that, in the opinion of the principal investigator, would interfere with the ability to adhere to study requirements.
5. History of myocardial infraction or angina.
6. Uncontrollable acute or chronic diseases, including hypertension or diabetes.
7. Second malignancy or cancer metastasis
8. HBV or HCV carrier
9. WBC below 4000 or ANC below 2000 on D1 of Cycle 1
10. Participation in investigational drug study within the past 30 days

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
% change from Visit 5 (C2, Day 1) to Visit 7 (C2, Day 15) in WBC, | % change from Visit 5 (C2, Day 1) to Visit 7 (C2, Day 15) in WBC,
% change from Visit 5 (C2, Day 1) to Visit 7 (C2, Day 15) in ANC | % change from Visit 5 (C2, Day 1) to Visit 7 (C2, Day 15) in WBC

SECONDARY OUTCOMES:
QOL analysis using EORTC questionnaires ndex scores | % change from Visit 5 (C2, Day 1) to Visit 7 (C2, Day 15) in QOL index scores
Inter-group comparison of Quality of Life survey collected for Cycle 2 | % change from Visit 5 (C2, Day 1) to Visit 7 (C2, Day 15) in QOL index scores
Within group analysis (based on "same person comparison"), on the change of WBC/ANC and QOL index scores | % change from Visit 5 (C2, Day 1) to Visit 7 (C2, Day 15) in QOL index scores

CONTACTS AND LOCATIONS:
Overall Officials: Tsu-Yi Chao, M.D, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Neihu, Taiwan